CLINICAL TRIAL: NCT04397484
Title: A Prospective Randomized Comparison of the Effects of Lidocaine and Levobupivacaine on Block Dynamics After a Subparaneural Popliteal Sciatic Nerve Block
Brief Title: Prospective RCT Lidocaine & Levobupivacaine on Block Dynamics After Subparaneural Popliteal Sciatic Nerve Block
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof Manoj K Karmakar, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020.127-T
Record Dates: First submitted 2020-05-13; First posted 2020-05-21 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Musculoskeletal Diseases or Conditions
Keywords: RCT; Lidocaine (Xylocaine) vs levobupivacaine; sciatic nerve block
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Levobupivacaine; Lidocaine; Epinephrine

STUDY DESIGN:
Intervention Model Description: The randomization sequence will be generated using online randomization software. The randomization sequence will be assigned as Group 1 =0.5% Chirocaine (levobupivacaine) and Group 2 =1.5% Xylocaine with adrenaline 1:200,000, and the group allocation will be sealed within an opague envelop by a research assistant, who is not involved in this study. After recruitment, patients will be randomly allocated to receive ultrasound guided subparaneural popliteal sciatic nerve block below bifurcation using either 0.5% Chirocaine (levobupivacaine) (Group 1) or 1.5% Xylocaine with adrenaline 1: 200,000 (Group 2).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 1. Patients will be blinded to the treatment arm in which he/she is allocated to.
  2. Anesthesiologist performing the block will receive identical syringes with equal volume of local anaesthetics, prepared by a nurse/ pharmacist who is not involved in the study.
  3. Anaesthesiologist performing the block will be blinded.
  4. Outcome assessor assessing the outcomes will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levobupivacaine (Active Comparator): 0.5% levobupivacaine (0.5% Chirocaine) 30ml (150mg) will be injected once for regional anaesthesia before surgery
  Interventions: Drug: 0.5% Levobupivacaine
- Xylocaine + adrenaline (Active Comparator): 2% Xylocaine with adrenaline 1:200,000 30ml (450mg) will be injected once for regional anaesthesia before surgery
  Interventions: Drug: 2% Xylocaine with adrenaline 1:200,000

INTERVENTIONS:
Drug: 0.5% Levobupivacaine — The plane where the sciatic nerve bifurcates will at first be identified by utlrasound. 22-gauge insulated nerve block needle will be inserted in the short axis (out-of-plane) of the ultrasound transducer, and advanced toward the cleavage between the common peroneal nerve and the tibial nerve, which is the easiest location for needle access into subparaneural compartment.Once the needle tip enters the subparaneural compartment 2-3 ml of normal saline will be injected (hydro-distension) to create a halo around both the common peroneal nerve and tibial nerve distally and the sciatic nerve proximally. The needle is then redirected to place its tip into the paraneural sheath of the common peroneal and tibial nerve through the same skin puncture and 15ml of study drug will be injected at each site (total 30ml).
  Other Names: Chirocaine
  Arms: Levobupivacaine
Drug: 2% Xylocaine with adrenaline 1:200,000 — The plane where the sciatic nerve bifurcates will at first be identified by utlrasound. 22-gauge insulated nerve block needle will be inserted in the short axis (out-of-plane) of the ultrasound transducer, and advanced toward the cleavage between the common peroneal nerve and the tibial nerve, which is the easiest location for needle access into subparaneural compartment.Once the needle tip enters the subparaneural compartment 2-3 ml of normal saline will be injected (hydro-distension) to create a halo around both the common peroneal nerve and tibial nerve distally and the sciatic nerve proximally. The needle is then redirected to place its tip into the paraneural sheath of the common peroneal and tibial nerve through the same skin puncture and 15ml of study drug will be injected at each site (total 30ml).
  Other Names: Lignocaine and Adrenaline; Lidocaine and Adrenaline
  Arms: Xylocaine + adrenaline

SUMMARY:
Sciatic nerve block at the popliteal fossa is indicated for foot or ankle surgery, and the introduction of ultrasound guidance (USG) has improved the ease and accuracy of the performance of this block. Recent studies proved that subparaneural injection is associated with faster block onset, higher block success rate, and prolonged block duration suggesting subparaneural compartment of the sciatic nerve is a desirable site for local anaesthetic injection. Data from an ongoing trial in the investigator's institution comparing the block dynamics of subparaneural injection of 30ml 0.5% levobupivacaine (Chirocaine) above and below the bifurcation of the sciatic nerve at popliteal fossa has also shown that the time to 'readiness for surgery' was faster when the injection was performed below the bifurcation of the sciatic nerve. Lidocaine (Xylocaine) has a better pharmacokinetic and pharmacodynamics profile than levobupivacaine and is also widely used as local anaesthetic agent in clinical practice. Since there is no data comparing the block dynamics of lidocaine and levobupivacaine, this study aims to study and compare the block dynamics of lidocaine and levobupivacaine when given as a subparaneural injection below the bifurcation of the sciatic nerve at the popliteal fossa. In this study, the investigator hypothesizes that the use of lidocaine as the sole agent for this block will fasten the time to 'readiness for surgery' as compared to levobupivacaine when given as a subparaneural injection below the bifurcation of the sciatic nerve at the popliteal fossa.

DETAILED DESCRIPTION:
This study will involve performing ultrasound guided subparaneural popliteal sciatic nerve block for 40 patients by using either Lidocaine or Levobupivacaine. Both are commonly used local anaesthetics for regional anaesthesia in daily clinical practice. Patients will be enrolled from the elective orthopaedic surgical list at Prince of Wales Hospital after informed consent.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III
* adult and scheduled to undergo elective forefoot surgery under regional anaesthesia

Exclusion Criteria:

* patient refusal
* ASA physical status > III
* pregnancy
* neuromuscular disorder
* prior surgery in the popliteal fossa
* coagulopathy
* allergy to local anaesthetic drugs
* skin infection at the site of needle insertion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Complete sensory blockade | assessed within the first 30 minutes
  Proportion of patients achieving complete sensory blockade (sensory score=0) at 30 minutes; Sensory score: VRS 0-100; 0=no sensation, 100=normal sensation

SECONDARY OUTCOMES:
Complete motor blockade | assessed within the first 50 minutes after nerve block at regular intervals (5min, 10min, 15min, 20min, 25min, 30min, 40min, 50min)
  Proportion of patients achieving complete motor blockade (motor score=0); Motor score: VRS 0-2; 2=normal, 1=paresis, 0=paralysis
Time to readiness for surgery | assessed within the first 50 minutes after nerve block at regular intervals (5min, 10min, 15min, 20min, 25min, 30min, 40min, 50min)
  Sensory score =<30 and motor score=<1
Time to complete sensory and motor block | assessed within the first 50 minutes after nerve block at regular intervals (5min, 10min, 15min, 20min, 25min, 30min, 40min, 50min)
  Sensory score =0 and motor score=0
Paresthesia | Intraoperative (during the period of undergoing the nerve block)
  Any incidence of paresthesia during the nerve block
complications | after the nerve block till the end of surgery
  Any complications during and right after the nerve block directly related to local anaesthetic toxicity
Discomfort score | assess once 1 day before surgery
  the degree of discomfort during the nerve block (NRS : 0-100; 0=no discomfort, 100 very uncomfortable)

CONTACTS AND LOCATIONS:
Overall Officials: Manoj K Karmakar, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No